CLINICAL TRIAL: NCT00719030
Title: A Randomized, Placebo-controlled, Pre-surgical Study of the Effects of Pomegranate Pills in Men With Prostate Cancer Prior to Radical Prostatectomy
Brief Title: A Study Of the Effectiveness Of Pomegranate Pills in Men With Prostate Cancer Before Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GUP-0515-02
Record Dates: First submitted 2008-07-15; First posted 2008-07-21 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pomegranate pill
  Interventions: Dietary Supplement: Pomegranate pill
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Pomegranate pill placebo

INTERVENTIONS:
Dietary Supplement: Pomegranate pill — Pomegranate extract pill
  Other Names: PomX
  Arms: 1
Dietary Supplement: Pomegranate pill placebo — Pomegranate pill placebo
  Other Names: POM-X placebo
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effects of pomegranate polyphenol pills (POM-X) and a placebo (sugar pill) on prostatic oxidative stress. The placebo is a pill that looks like the POM-X pill but does not have an active ingredient.

DETAILED DESCRIPTION:
Subjects will receive POM-X or placebo pills daily for up to 4 weeks prior to undergoing radical prostatectomy for prostate cancer. Biomarkers in the blood, urine, and prostate tissue will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate, without evidence of spread beyond to lymph nodes, bone, or visceral organs.
2. Radical prostatectomy scheduled at Duke or Johns Hopkins.
3. Initial prostate biopsy available for review with tumor involving 2 or more core biopsies based on pathologic review.
4. Age ≥ 18 years of age.
5. Willingness and ability to sign an informed consent document.
6. Agreement with complete abstinence from other commercially available pomegranate products during the course of the study.
7. No prior allergy to pomegranate dietary agents.
8. No significant medical or psychiatric condition that would make the patient a poor protocol candidate.
9. The patient agrees to stop taking dietary or vitamin supplements (lycopene, vitamin E, selenium, genistein) or herbal supplements (eg. saw palmetto) for 2-weeks prior to staring the study.
10. The patient is not taking LHRH agonists, androgen receptor blocking agents or finasteride, and has not undergone bilateral orchiectomy.
11. Patient has not received experimental medications within the past six months.

Exclusion Criteria:

1. Significant concomitant medical or psychiatric condition that, in the opinion of the investigator, would make the participant a poor protocol candidate.
2. Concomitant or antecedent hormonal therapy.
3. Known allergy to pomegranate juice.
4. Subjects unable or unwilling to comply with protocol requirements.
5. Evidence of metastatic disease on physical examination or on CT or bone scan.
6. Use of finasteride, dutasteride at any point during the study.
7. Clinically significant abnormal laboratory value >2X the upper limit of normal (2XULN).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pomegranate oxidative stress | On day of prostate surgery following 4 weeks of taking POM-X or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Allan J Pantuck, MD, Principal Investigator — University of California, Los Angeles; Michael Carducci, MD, Principal Investigator — Johns Hopkins Medical Center; Stephen J Freedland, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - UCLA, Los Angeles, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina